CLINICAL TRIAL: NCT05433584
Title: A Randomized, Open-Label, Parallel-Group, Two-Arm, Phase 4 Study to Evaluate the Long-Term Efficacy and Safety of Tirzepatide Compared With Intensified Conventional Care in Adults When Initiating Treatment Early in the Course of Type 2 Diabetes
Brief Title: A Study of Tirzepatide Compared With Intensified Conventional Care in Adult Participants With Type 2 Diabetes
Acronym: SURPASS-EARLY
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17205; I8F-MC-GPHE (Other: Eli Lilly and Company); 2022-000130-42 (EudraCT Number); 2022-5010733-40-00 (Other: EU Trial Number); U1111-1282-0263 (Registry Identifier: World Health Organization)
Record Dates: First submitted 2022-06-22; First posted 2022-06-27 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes
Keywords: T2D; Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Tirzepatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tirzepatide (Experimental): Participants will receive tirzepatide at the maximum tolerated dose subcutaneously (SC)
  Interventions: Drug: Tirzepatide
- Intensified Conventional Care Dose (Active Comparator): Participants will receive an antihyperglycemic medication
  Interventions: Drug: Antihyperglycemic medication

INTERVENTIONS:
Drug: Tirzepatide — Administered SC
  Other Names: LY3298176
  Arms: Tirzepatide
Drug: Antihyperglycemic medication — As prescribed
  Arms: Intensified Conventional Care Dose

SUMMARY:
This study aims to investigate the efficacy and safety of tirzepatide in participants with type 2 diabetes (T2D) compared to other existing treatment options when treatment is initiated early.

ELIGIBILITY:
Inclusion Criteria:

* Have, within the last 4 years, been diagnosed with T2D based on the World Health Organization classification or other locally applicable diagnostic standards.
* Have HbA1c ≥7% to ≤9.5% as determined by the central laboratory.
* Have been on a stable treatment of metformin only at least 90 days preceding baseline

  * with the minimum effective dose of ≥1500 mg/day, but not higher than the maximum approved dose per country-specific label, or
  * <1500 mg/day in case of intolerance of full therapeutic dose.

Exclusion Criteria:

* Have type 1 diabetes mellitus
* Have a history of chronic or acute pancreatitis any time prior to study entry
* Have a history of

  * proliferative diabetic retinopathy
  * diabetic macular edema, or
  * no proliferative diabetic retinopathy requiring immediate or urgent treatment
* Are at high risk for cardiovascular disease (CVD) in the investigator's opinion or have a history of any of these CV conditions prior to study entry

  * myocardial infarction
  * percutaneous coronary revascularization procedure
  * carotid stenting or surgical revascularization
  * nontraumatic amputation
  * peripheral vascular procedure (e.g., stenting or surgical revascularization)
  * cerebrovascular accident (stroke), or congestive heart failure
* Have family or personal history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2 (MEN2)
* Have within 90 days prior to screening received treatment with medications intended to promote weight loss. This includes prescribed, over the counter, or alternative remedies
* Have an estimated glomerular filtration rate (eGFR) <30 mL/minute/1.73 m2 (or lower than the country-specific threshold for discontinuing metformin therapy per local label), calculated by chronic kidney disease-epidemiology equation as determined by central laboratory at screening.
* Have been treated with any injectable glucagon-like peptide-1 (GLP-1) receptor agonists and insulin prior to screening.

  * Exception: use of insulin for gestational diabetes or short-term use (<14 days) for acute conditions such as acute illness, hospitalization, or elective surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 780 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-10-21 (Actual); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Hemoglobin A1c (HbA1c) | Baseline, Week 104

SECONDARY OUTCOMES:
Change from Baseline in HbA1c | Baseline, Week 208
Change from Baseline in Weight | Baseline, Week 104
Change from Baseline in Weight | Baseline, Week 208
Change from Baseline in Waist Circumference | Baseline, Week 104
Change from Baseline in Waist Circumference | Baseline, Week 208
Change from Baseline in Fasting Serum Glucose (FSG) | Baseline, Week 104
Change from Baseline in FSG | Baseline, Week 208
Change from Baseline in Lipids | Baseline, Week 104
Change from Baseline in Lipids | Baseline, Week 208
Percentage of Participants Achieving HbA1c <7.0% | Week 104
Percentage of Participants Achieving HbA1c ≤6.5% | Week 104
Percentage of Participants Achieving HbA1c <5.7% | Week 104
Percentage of Participants Achieving HbA1c <7.0% | Week 208
Percentage of Participants Achieving HbA1c ≤6.5% | Week 208
Percentage of Participants Achieving HbA1c <5.7% | Week 208
Change from Baseline in Weight loss of ≥5%, | Baseline, Week 104
Change from Baseline in Weight loss of ≥10% | Baseline, Week 104
Change from Baseline in Weight loss of ≥15% | Baseline, Week 104
Change from Baseline in Weight loss of ≥5% | Baseline, Week 208
Change from Baseline in Weight loss of ≥10% | Baseline, Week 208
Change from Baseline in Weight loss of ≥15% | Baseline, Week 208
A Composite Endpoint of HbA1c, Weight loss and Hypoglycemia | Week 104
  A composite endpoint defined as HbA1c ≤ 6.5%, weight loss ≥10%, no hypoglycemia, defined as blood glucose (BG) <54 milligram/deciliter (mg/dL) <3.0 millimole/liter (mmol/L) and/or severe hypoglycemia
A Composite Endpoint of HbA1c, Weight loss and Hypoglycemia | Week 208
  A composite endpoint defined as HbA1c ≤ 6.5%, weight loss ≥10%, no hypoglycemia, defined as BG <54 mg/dL (<3.0 mmol/L) and/or severe hypoglycemia
Change from Baseline in β-cell Glucose Sensitivity | Baseline, Week 104
  β-cell Glucose Sensitivity assessed by Oral Glucose Tolerance Test (OGTT)
Change from Baseline in β-cell glucose sensitivity | Baseline, Week 208
  Change from baseline in β-cell glucose sensitivity assessed by OGTT
Change from Baseline in Insulin Secretion Rate at a Fixed Glucose Concentration | Baseline, Week 104
  Insulin Secretion Rate assessed by OGTT
Change from Baseline in Insulin Secretion Rate at a Fixed Glucose Concentration | Baseline, Week 208
  Insulin Secretion Rate assessed by OGTT
Change from Baseline in Postprandial Insulin Sensitivity Indices | Baseline, Week 104
  Postprandial Insulin Sensitivity Indices assessed by OGTT
Change from Baseline in Postprandial Insulin Sensitivity Indices | Baseline, Week 208
  Postprandial Insulin Sensitivity Indices assessed by OGTT
Change from Baseline in Fasting and Post-challenge Glucose [total and incremental AUC(₀-₂₄₀min)] | Baseline through Week 104
  Fasting and Post-challenge Glucose [total and incremental AUC(₀-₂₄₀min)] assessed by OGTT
Change from Baseline in Fasting and Post-challenge Glucose [total and incremental (AUC₀-₂₄₀min)] | Baseline through Week 208
  Fasting and Post-challenge Glucose [total and incremental AUC(₀-₂₄₀min)] assessed by OGTT
Change from Baseline in the Impact of Weight on Quality of Life-Lite Clinical Trials Version (IWQOL-Lite-CT) - Physical Functioning Domain | Baseline, Week 104
Change from Baseline in the IWQOL-Lite-CT - Physical Functioning Domain | Baseline, Week 208

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (90):
- United States (32):
  - Cahaba Research - Trussville, Birmingham, Alabama
  - San Fernando Valley Health Institute, Canoga Park, California
  - Velocity Clinical Research, Huntington Park, Huntington Park, California
  - Velocity Clinical Research, San Diego, La Mesa, California
  - Clinical Trials Research, Lincoln, California
  - Velocity Clinical Research, Westlake, Los Angeles, California
  - Catalina Research Institute, LLC, Montclair, California
  - Velocity Clinical Research, North Hollywood, North Hollywood, California
  - Velocity Clinical Research, Panorama City, Panorama City, California
  - Western University of Health Sciences, Pomona, California
  - Velocity Clinical Research, Santa Ana, Santa Ana, California
  - New England Research Associates, LLC, Bridgeport, Connecticut
  - Excel Medical Clinical Trials, Boca Raton, Florida
  - Alliance for Multispecialty Research, LLC, Coral Gables, Florida
  - South Florida Clinical Research Institute, Margate, Florida
  - Emory University School of Medicine- Grady Campus, Atlanta, Georgia
  - Center for Advanced Research & Education, Gainesville, Georgia
  - Qualmedica Research, LLC, Evansville, Indiana
  - Iowa Diabetes and Endocrinology Research Center, West Des Moines, Iowa
  - Qualmedica Research, Bowling Green, Kentucky
  - NECCR PrimaCare Research, Fall River, Massachusetts
  - SKY Integrative Medical Center/SKYCRNG, Ridgeland, Mississippi
  - StudyMetrix Research, City of Saint Peters, Missouri
  - Clinvest Research LLC, Springfield, Missouri
  - Research Foundation of SUNY - University of Buffalo, Buffalo, New York
  - Lucas Research, Inc, Morehead City, North Carolina
  - The Corvallis Clinic, P.C., Corvallis, Oregon
  - Clinical Research of Philadelphia, Philadelphia, Pennsylvania
  - Preferred Primary Care Physicians, Uniontown, Pennsylvania
  - Tribe Clinical Research, LLC, Greenville, South Carolina
  - Velocity Clinical Research, Spartanburg, Spartanburg, South Carolina
  - Dallas Diabetes Research Center, Dallas, Texas
- Argentina (5):
  - Centro de Investigaciones Metabólicas (CINME), Ciudad Autónoma de Buenos Aire, Buenos Aires
  - Instituto de Investigaciones Clínicas Mar del Plata, Mar del Plata, Buenos Aires
  - Go Centro Medico San Nicolás, San Nicolás de los Arroyos, Buenos Aires
  - CIAD Moron, Morón, Buenos Air
  - Centro Médico Viamonte, Buenos Aires, Ciudad Aut
- Canada (4):
  - Dr. M.B. Jones Inc., Victoria, British Columbia
  - Bluewater Clinical Research Group Inc., Sarnia, Ontario
  - Stouffville Medical Centre, Stouffville, Ontario
  - 9109-0126 Quebec Inc., Montreal, Quebec
- Germany (8):
  - ClinPhenomics CVC GmbH, Frankfurt am Main, Hesse
  - Diabetes- und Stoffwechselpraxis Bochum, Bochum, North Rhine-Westphalia
  - InnoDiab Forschung Gmbh, Essen, North Rhine-Westphalia
  - Zentrum für klinische Studien, Saint Ingbert, Saarland
  - Arztpraxis Christine Kosch Pirna, Pirna, Saxony
  - RED-Institut GmbH, Oldenburg in Holstein, Schleswig-Holstein
  - Diabetespraxis Mergentheim, Bad Mergentheim
  - Diabetes Zentrum Dr. Tews, Gelnhausen
- Israel (9):
  - Edith Wolfson Medical Center, Holon, Central District
  - Rabin Medical Center, Petah Tikva, Central District
  - Sheba Medical Center, Ramat Gan, Central District
  - Kaplan Medical Center, Rehovot, Central District
  - Hadassah Medical Center, Jerusalem, Jerusalem
  - Bnai Zion Medical Center, Haifa, Northern District
  - Clalit Health Services - Sakhnin Community Clinic, Sakhnin, Northern District
  - Clalit Health Services - Atlit, Atlit, Southern District
  - Linn Medical Center, Haifa, Ḥeifā
- Italy (8):
  - A.O.U.C. Policlinico di Bari, Bari, Apulia
  - University of Naples Federico II, Napoli, Campania
  - Centro Cardiologico Monzino, Milan, Milano
  - Ospedale Civile Santa Croce Pronto Soccorso, Moncalieri, Piedmont
  - Ospedale san Giovanni di Dio-Diabetologia, Olbia, Sardinia
  - A.O.U. Policlinico Paolo Giaccone, Palermo, Sicily
  - Azienda Ospedaliera Universitaria Pisana, Pisa, Tuscany
  - AOU Renato Dulbecco, Catanzaro
- Mexico (3):
  - Private Practice - Dr. Arechavaleta Granell Maria del Rosario, Guadalajara, Jalisco
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Monterrey, Nuevo León
  - Investigacion En Salud Y Metabolismo Sc, Chihuahua City
- Puerto Rico (3):
  - San Juan Bautista School of Medicine - Clinical Research Unit, Caguas, PR
  - GCM Medical Group, PSC - Hato Rey Site, San Juan, PR
  - Dorado Medical Complex, Dorado
- Romania (7):
  - Diabdana, Oradea, Bihor County
  - C.M.D.T.A. Neomed, Brasov, Brașov County
  - Centrul Medical NutriLife, Bucharest, București
  - Gama Diamed, Mangalia, Constanța County
  - Diabmed Dr. Popescu Alexandrina, Ploieşti, Prahova
  - Milena Sante, Galați
  - Clinica Korall, Satu Mare
- Slovakia (4):
  - MEDIKALS, Piešťany
  - ProDia s.r.o., Považská Bystrica
  - JAL, Trnava
  - IRIDIA, Vrútky, Žilina Region
- United Kingdom (7):
  - Aberdeen Royal Infirmary, Aberdeen, Aberdeen City
  - Ninewells Hospital and Medical School, Dundee, Angus
  - Staploe Medical Centre, Ely, Cambridgeshire
  - Knowle House Surgery, Plymouth, Devon
  - Hull Royal Infirmary, Hull, Kingston Upon Hull
  - Leicester General Hospital, Leicester, Leicestershire
  - Wickersley Health Centre - Clifton Medical Centre, Rotherham

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- See also: A Study of Tirzepatide Compared With Intensified Conventional Care in Adult Participants With Type 2 Diabetes (SURPASS-EARLY) — https://trials.lillytrialguide.com/en-US/trial/6uDOXjWupVuV6MjrZKbsNy